CLINICAL TRIAL: NCT05154214
Title: Prospective Study of Surgical Treatment of Children With Obstructive Sleep Apnea and Small Tonsils or Down Syndrome
Brief Title: Surgical Treatment of Children With OSA and Small Tonsils or Down Syndrome
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Derek Lam, MD, MPH, Principal Investigator, Oregon Health and Science University
Other Study IDs: STUDY00023287
Record Dates: First submitted 2021-11-15; First posted 2021-12-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea of Child
Keywords: Adenotonsillectomy; Drug-induced sleep endoscopy; pediatric; otolaryngology; OSA; sleep apnea; Down Syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes; Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adenotonsillectomy: Excision of the palatine tonsils and excision or ablation of the adenoids by each individual surgeon's preferred techniques.
  Interventions: Procedure: Adenotonsillectomy
- Drug-induced sleep endoscopy directed surgery (DISE): DISE will be performed by the surgeon performing the surgical intervention. The DISE Rating Scale assesses the degree of maximal closure or obstruction at six locations in the upper airway: the nose, nasopharynx (adenoids), velopharynx (soft palate), oropharynx (tonsils), tongue base (tongue, lingual tonsils), and larynx (epiglottis, arytenoids). The degree of obstruction is scored on a 3-point rating scale as none (0), partial (+1), or complete (+2) at each anatomic site. The rating at each anatomic level can be summed into a DISE Rating Scale total. The actual surgery performed will determine which established surgical treatments will be used based on the results of the DISE.
  Interventions: Procedure: Drug-induced sleep endoscopy directed surgery

INTERVENTIONS:
Procedure: Adenotonsillectomy — Removal of tonsils and adenoids
  Groups: Adenotonsillectomy
Procedure: Drug-induced sleep endoscopy directed surgery — Surgeries selected based on direct visualization of airway collapse using endoscopy during drug-induced sleep
  Groups: Drug-induced sleep endoscopy directed surgery (DISE)

SUMMARY:
The purpose of this study is to prospectively compare the effectiveness of a novel personalized approach to the surgical treatment of obstructive sleep apnea (OSA) in children, drug induced sleep endoscopy (DISE) directed surgery versus the standard adenotonsillectomy (AT). This will also serve to test the feasibility of recruiting families for a future randomized protocol comparing the same surgical techniques. It is the investigators' central hypothesis that a personalized DISE-directed surgical approach that uses existing procedures to address the specific fixed and dynamic anatomic features causing obstruction (ie, anatomic endotypes) in each child with small tonsils or Down syndrome will be superior to the currently recommended standard first line approach of AT. This novel approach may improve OSA outcomes and reduce the burden of unnecessary AT or secondary surgery for persistent OSA after an ineffective AT. To test this hypothesis, the investigators will study children aged 2 to 18 years with clinically small tonsils (Brodsky score 1+ or 2+ on a scale 1+ to 4+) OR Down syndrome.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is defined as repetitive obstruction of the upper airway during sleep and has been estimated to affect 1-6% of the general pediatric population. Untreated OSA in children has been associated with childhood hypertension, autonomic dysfunction, attention-deficit/hyperactivity disorder, neurobehavioral impairment, and poor quality of life. These sequelae contribute to a 226% increase in health care utilization among children with OSA compared to controls, primarily in the form of increased hospitalizations, emergency department visits, and medication use. Adenotonsillar hypertrophy is considered the most common risk factor for OSA in children, and adenotonsillectomy (AT) is the first line treatment.

Although AT is the recommended first line treatment for pediatric OSA in treatment guidelines, multiple studies have demonstrated that AT is not always curative, with estimates of persistent OSA after AT ranging from 25 to 75%. Many risk factors for AT failure have been reported, but the impact of tonsil size on AT outcome remains a controversial topic. Not every child with enlarged tonsils will have OSA, and conversely, there are many children with proven OSA who do not have clinically large tonsils or adenoids. The prevalence of small tonsils (1+ or 2+ on Brodsky tonsil scoring scale of 1+ to 4+) has been reported to be 67-70% among children with symptoms of OSA presenting to either the emergency department or a pediatric pulmonology clinic. Clinic assessment of tonsil size during an awake examination has not consistently correlated with either baseline disease severity or response to AT. The outcome of AT in children with small tonsils (Brodsky 1+ or 2+) remains unknown and clinical decisions in children with small tonsils are not evidence-based.

Patients with Down Syndrome have a higher incidence of OSA than the general pediatric population, with rates of 30-60%, resulting in increased morbidity and decreased quality of life for affected individuals. Children with Down Syndrome often undergo T&A for obstructive sleep apnea; however 30-50% will have persistent obstructive sleep patterns requiring continuous positive pressure airway support (CPAP) or tracheotomy. Persistent obstruction is attributed to anatomic and physiologic differences in this population, including reduced muscular tone, macroglossia, maxillary hypoplasia, and lingual tonsil hypertrophy.

Drug-induced sleep endoscopy (DISE) enables direct observation of the sites and patterns of obstruction during sedated sleep. DISE increasingly helps guide surgical decision-making in adult OSA, and the investigators hypothesize DISE can guide surgical decisions in pediatric OSA and improve outcomes. Towards that end, the study team has developed and validated the DISE Rating Scale in children. Furthermore, the investigators have demonstrated DISE ratings of adenotonsillar obstruction during sedated sleep are strongly associated with both OSA severity and response to AT, unlike clinic assessments of tonsil size. This preliminary data and others' studies have identified non-adenotonsillar obstruction can also occur at the nose, palate, base of tongue, and larynx. DISE findings in surgically naïve children and the outcomes of procedures based on those findings have been reported in mostly small observational case series. The surgical plan may be modified from the standard AT in up to 77% of children based on DISE findings. These alternative procedures can be less invasive (e.g., only isolated adenoidectomy or isolated tonsillectomy) or include procedures to address other anatomic sites in addition to or instead of the tonsils and adenoids. The most commonly reported non-adenotonsillar sites of obstruction are the nose, velopharynx (soft palate), tongue base, and the larynx. DISE-directed surgery at these sites may improve pediatric OSA outcomes, but existing studies are small, uncontrolled case series in heterogeneous study populations. There are no trials directly comparing AT and DISE-directed surgery in the common scenario of surgically naïve children with small tonsils. This study will inform a future randomized trial that has the potential to change the paradigm of treating OSA in children with small tonsils or Down syndrome, thereby improving outcomes, and reducing inappropriate AT and need for secondary sleep surgery.

ELIGIBILITY:
Inclusion Criteria:

* Moderate OSA (oAHI ≥ 5),
* Clinically small tonsils (Brodsky score 1+ or 2+) AND/OR Down syndrome
* Desiring surgical treatment.
* English or Spanish speaking

Exclusion Criteria:

* Non-Down Syndrome neuromuscular disorder, craniofacial anomaly, genetic abnormality, subglottic or tracheal stenosis, tracheostomy dependence.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited from the Oregon Health and Science University pediatric otolaryngology clinic and from the pediatric sleep medicine clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Change in Pediatric Quality of Life (PedsQL), a generic quality of life scale | 6 months post-surgery
  Parent and child-reported surveys, higher scores indicate better quality of life, mean scores 0-100
Parent-reported ease of participation | 6 months post-surgery
  Parent-reported survey or parent interview
Parent-reported barriers to recruitment | Initial visit
  Parent-reported survey or parent interview
Change in Obstructive Sleep Apnea -18 (OSA-18): disease-specific quality of life survey | 6 months post-surgery
  Parent-reported survey, higher scores mean higher disease burden, scores from 18-126
Parent-reported barriers to recruitment | 6 months post-surgery
  Parent-reported survey or parent interview

SECONDARY OUTCOMES:
Change in Obstructive Apnea-Hypopnea Index (oAHI) | 6 months post-surgery
  As measured in clinical polysomnography (PSG)
Change in Total Apnea-Hypopnea Index | 6 months post-surgery
  As measured in clinical polysomnography (PSG)
Change in REM Apnea-Hypopnea Index (REM AHI) | 6 months post-surgery
  As measured in clinical polysomnography (PSG)
Change in Minimum Oxygen Saturation (Min SpO2) | 6 months post-surgery
  As measured in clinical polysomnography (PSG)
Change in Mean End Tidal CO2 (ETCO2) | 6 months post-surgery
  As measured in clinical polysomnography (PSG)
Change in Max End Tidal CO2 (ETCO2) | 6 months post-surgery
  As measured in clinical polysomnography (PSG)
Change in Oxyhemoglobin desaturation ≥3% Index (ODI) | 6 months post-surgery
  As measured in clinical polysomnography (PSG)
Change in % Total Sleep Time with ETCO2 > 45/50 mmHg | 6 months post-surgery
  As measured in clinical polysomnography (PSG)

CONTACTS AND LOCATIONS:
Overall Officials: Derek J Lam, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No